CLINICAL TRIAL: NCT03391947
Title: Comparison of a Semilunar Coronally Positioned Flap and Conventional Coronally Advanced Flap for the Treatment of Gingival Recession- A Split-mouth, Randomized Prospective Comparative Controlled Clinical Trial
Brief Title: Semilunar and Conventional Coronally Positioned Flap for the Treatment Gingival Recession
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Perio-01-2018
Record Dates: First submitted 2017-12-31; First posted 2018-01-05 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Gingival Recession; Root Coverage
Keywords: gingival recession; semilunar coronally flap; coronally advanced flap
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Intervention Model Description: Split-mouth design, i.e. the right side will receive the first intervention, whereas the other side (the left side) will receive the second intervention.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- semilunar coronally positioned flap (Experimental): A semilunar incision will be done following the curvature of the gingival margin and ending about 2 to 3 mm short of the tip of the papillae. The most apical distance of this incision to the gingival margin will be obtained by adding the bone sounding measurement to the recession height. Perform a split-thickness dissection coronally from the incision, and connect it to an intrasulcular incision. The tissue will be collapsed coronally, covering the denuded root. The coronally repositioned gingival margin will be stabilized by coronally anchored suture with composite stops on the buccal surface of the tooth using flowable composite. Finally, the area will be covered with a periodontal dressing. This is called semilunar coronally positioned flap.
  Interventions: Procedure: semilunar coronally positioned flap
- coronally advanced flap (Active Comparator): Coronally positioned flap will be initiated with two vertical incisions, extending from a mesial and distal linear angle at the cementoenamel junction (CEJ) and go beyond the mucogingival junction. A split thickness flap will be prepared by sharp dissection mesial and distal to the recession and connected with an intra crevicular incision. On the facial aspect of the tooth, a full thickness flap, approximately 3-4 mm apical to crest of alveolar bone. Then, the flap will be returned and sutured it at 1 mm coronal to the CEJ after de-epithelize the papillae. The coronally repositioned gingival margin will be stabilized by coronally anchored suture with composite stops on the buccal surface of the tooth using flowable composite and sutured in the papilla region and releasing incision. Finally, the area will be covered with a periodontal dressing.
  Interventions: Procedure: coronally advanced flap

INTERVENTIONS:
Procedure: semilunar coronally positioned flap — The description of this intervention has been already given before
  Arms: semilunar coronally positioned flap
Procedure: coronally advanced flap — The description of this intervention has been already given before
  Arms: coronally advanced flap

SUMMARY:
A clinical evaluation of using the semilunar coronally position flap (SCPF) compared to the conventional coronally advanced flap (CAF) with modification to treat class I Miller gingival recession. The coronally repositioned gingival margin will be stabilized by coronally anchored suture with composite stops on the buccal surface of the tooth using flowable composite. The sample size will be ten patients. Each patient has bilateral Miller Class I gingival recessions; one will be treated with SCPF, while the other will be treated with CAF

DETAILED DESCRIPTION:
The aim of this study is to clinically compare between the semilunar coronally positioned flap (SCPF) and the conventional coronally advanced flap (CAF) after applying modification in both techniques to treat class I Miller gingival recession. Coronally repositioned gingival margin will be stabilized by coronally anchored suture with composite stops on the buccal surface of tooth using flowable composite for the treatment of gingival recession. Ten patients who have bilateral maxillary buccal Miller Class I gingival recession defects will be enrolled in this study. These defects will be distributed randomly into two groups: the test group (SCPF) and control group (CAF). Clinical parameters will be evaluated: visible plaque index (VPI), sulcus bleeding index (SBI), probing depth (PD), gingival recession height (GRH), gingival recession width (GRW), clinical attachment level (CAL), width of keratinized tissue (WKT), thickness of keratinized tissue (TKT), change in the position of muco-gingival junction, vestibular depth, wound healing index (WHI), the percentage of root coverage (RC) and root coverage esthetic score (RES) system. A questionnaire will be given to each patient, which includes evaluation of the pain intensity, root sensitivity, and satisfaction with aesthetic by using the visual analog scale (VAS) and questions about the number of analgesic pills consumed per day.

ELIGIBILITY:
Inclusion Criteria:

* Patients are in general good health.
* The patient is non-smoker (less than 10 cigarettes per day) and non-alcoholic.
* Female participants must not be pregnant and not at menstrual period during surgery.
* The patient is committed to the oral care, and has a healthy periodontium.
* Absence of severe oral habits.
* They have not taken medication known to interfere with periodontal tissue health or healing in the preceding 6 months.
* Presence of bilateral buccal Miller class I gingival recessions (≤5 mm) in maxillary incisors, canines, or premolars.
* Presence width of keratinized tissue (WKT) ≥2 mm.
* The tooth is vital and absence of caries or restorations in the areas that will be treated.
* Pocket depth less than 3 mm without bleeding on probing (BOP).

Exclusion Criteria:

1. Patients less than 18 years old
2. Patients with untreated periodontal disease.
3. Smokers.
4. Immunosuppressive systemic diseases (like cancer, AIDS, diabetes…)
5. Miller's class II, III or IV gingival recession defects.
6. Presence of apical radiolucency or root surface restoration or caries at the defect site
7. Medications influence on the health of the gingival tissue (like calcium channel blockers, immunosuppressive systemic diseases (like cancer, AIDS, diabetes…) or Long-term steroid use

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-12-20 (Actual)

PRIMARY OUTCOMES:
Change in the amount of root coverage | (1) one day before the surgery, (2) at 2 weeks post-surgery, (3) at 1 month post-surgery, (4) and at 3 months post-surgery
  this will be measured as a change of gingival recession height GRH (the distance from the cemento-enamel junction CEJ to the gingival margin GM by using an endodontic finger spreader attached to a rubber stopper and after removing the spreader, penetration depth was measured with a caliper of 0.01-mm resolution) from baseline and follow-up period.

SECONDARY OUTCOMES:
Change in visible plaque index | (1) one day before the surgery, (2) at 2 weeks post-surgery, (3) at 1 month post-surgery, (4) and at 3 months post-surgery
  Score 0 - No plaque Score 1 - Separate flecks of plaque at the cervical margin of the tooth Score 2 - A thin continuous band of plaque at the cervical margin of the tooth Score 3 - A band of plaque wider then 1mm covering less than 1/3rd of the crown of the tooth Score 4 - Plaque covering at least 1/3rd but less than 2/3rd of the crown of the tooth Score 5 - Plaque covering 2/3rd or more of the crown of the tooth
Change in sulcus bleeding index | (1) one day before the surgery, (2) and at 3 months post-surgery
  will be evaluated visually (using an UNC-15 mm "University of North Carolina" periodontal probe) Score 0 - health looking papillary and marginal gingiva no bleeding on probing; Score 1 - healthy looking gingiva, bleeding on probing; Score 2 - bleeding on probing, change in color, no edema; Score 3 - bleeding on probing, change in color, slight edema; Score 4 -bleeding on probing, change in color, obvious edema; Score 5 -spontaneous bleeding, change in color, marked edema
Change in probing depth | (1) one day before the surgery, (2) and at 3 months post-surgery
  Probing depth will be measured as the distance from the gingival margin GM to the bottom of the gingival sulcus by using a periodontal probe (UNC 15 "University of North Carolina") with a rubber stopper.
Change in the clinical attachment level | (1) one day before the surgery, (2) and at 3 months post-surgery
  clinical attachment level will be calculated as the sum of the gingival recession height and the probing depth (mentioned above).
Change in the gingival recession width | (1) one day before the surgery, (2) at 2 weeks post-surgery, (3) at 1 month post-surgery, (4) and at 3 months post-surgery
  Gingival recession width will be measured from one border of the recession to another at the CEJ by using an endodontic finger spreader attached to a rubber stopper and after removing the spreader, penetration depth was measured with a caliper of 0.01-mm resolution
Change in the width of keratinized tissue | (1) one day before the surgery, (2) at 2 weeks post-surgery, (3) at 1 month post-surgery, (4) and at 3 months post-surgery
  The width of the keratinized tissue will be measured as the distance between the most apical point of the GM and the MGJ by using an endodontic finger spreader attached to a rubber stopper and after removing the spreader, penetration depth was measured with a caliper of 0.01-mm resolution.
Change in the thickness of the keratinized tissue | (1) one day before the surgery, (2) and at 3 months post-surgery
Change in the position of the mucogingival junction | (1) one day before the surgery, (2) at 2 weeks post-surgery, (3) at 1 month post-surgery, (4) and at 3 months post-surgery
  The distance between the incisal edge and the mucogingival junction will be measured using an endodontic finger spreader attached to a rubber stopper and after removing the spreader, penetration depth was measured with a caliper of 0.01-mm resolution
Change in the wound healing index | (1) at two weeks following surgery and (2) at one month following surgery.
  Wound healing index will be recorded after surgery using the following criteria:
  score 1 = uneventful healing with no gingival edema, erythema, suppuration, patient discomfort, or flap dehiscence score 2 = uneventful healing with slight gingival edema, erythema, patient discomfort, or flap dehiscence, but no suppuration score 3 = poor wound healing with significant gingival edema, erythema, patient discomfort, flap dehiscence, or any suppuration
Change in post-operative pain level | at 2 hours, 24 hours, 48 hours, 72 hours following surgery and at 1-week after surgery
  Using a 10 cm-visual analog scale
Patients' satisfaction with aesthetics | at three months post-surgery
  Using a 10 cm-visual analog scale (VAS), patients' satisfaction with the aesthetic result will be recorded with 0 indicating very bad, 5 indicating average feelings and 10 indicating excellent result.
Change in root sensitivity | (1) one day before the surgery, (2) at 2 weeks post-surgery, (3) at 1 month post-surgery, (4) and at 3 months post-surgery
  Using a 10 cm-visual analog scale (VAS), patients' perception of root sensitivity will be recorded with zero indicating no pain or sensitivity, 5 indicating moderate pain or sensitivity and 10 indicating worst pain or sensitivity possible.

CONTACTS AND LOCATIONS:
Overall Officials: Hala Mohammad Walid Hala Mohammad Walid, DDS, Principal Investigator — MSc student in Periodontics, Periodontology Department, University of Damascus Dental School; Suleiman Dayoub, DDS MSc PhD, Study Chair — Professor of Periodontics, Department of Periodontology, University of Damascus Dental School
Locations (1):
- Department of Periodontics, University of Damascus Dental School, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Santana RB, Mattos CM, Dibart S. A clinical comparison of two flap designs for coronal advancement of the gingival margin: semilunar versus coronally advanced flap. J Clin Periodontol. 2010 Jul;37(7):651-8. doi: 10.1111/j.1600-051X.2010.01582.x. Epub 2010 Jun 1. PMID 20528963
- [Background] Bittencourt S, Del Peloso Ribeiro E, Sallum EA, Sallum AW, Nociti FH Jr, Casati MZ. Comparative 6-month clinical study of a semilunar coronally positioned flap and subepithelial connective tissue graft for the treatment of gingival recession. J Periodontol. 2006 Feb;77(2):174-81. doi: 10.1902/jop.2006.050114. PMID 16460241
- [Background] Bittencourt S, Ribeiro Edel P, Sallum EA, Sallum AW, Nociti FH Jr, Casati MZ. Root surface biomodification with EDTA for the treatment of gingival recession with a semilunar coronally repositioned flap. J Periodontol. 2007 Sep;78(9):1695-701. doi: 10.1902/jop.2007.060507. PMID 17760538
- [Background] Bhandari R, Uppal RS, Kahlon KS. Comparison of semilunar coronally advanced flap alone and in combination with button technique in the treatment of Miller's Class I and II gingival recessions: A pilot study. Indian J Dent Res. 2015 Nov-Dec;26(6):609-12. doi: 10.4103/0970-9290.176925. PMID 26888240
- [Background] Bittencourt S, Ribeiro Edel P, Sallum EA, Sallum AW, Nociti FH, Casati MZ. Semilunar coronally positioned flap or subepithelial connective tissue graft for the treatment of gingival recession: a 30-month follow-up study. J Periodontol. 2009 Jul;80(7):1076-82. doi: 10.1902/jop.2009.080498. PMID 19563287
- [Background] Ozcelik O, Haytac MC, Seydaoglu G. Treatment of multiple gingival recessions using a coronally advanced flap procedure combined with button application. J Clin Periodontol. 2011 Jun;38(6):572-80. doi: 10.1111/j.1600-051X.2011.01724.x. Epub 2011 Mar 28. PMID 21443557
- [Background] Kaval B, Renaud DE, Scott DA, Buduneli N. The role of smoking and gingival crevicular fluid markers on coronally advanced flap outcomes. J Periodontol. 2014 Mar;85(3):395-405. doi: 10.1902/jop.2013.120685. Epub 2013 May 31. PMID 23725027
- [Background] Pini-Prato G, Baldi C, Pagliaro U, Nieri M, Saletta D, Rotundo R, Cortellini P. Coronally advanced flap procedure for root coverage. Treatment of root surface: root planning versus polishing. J Periodontol. 1999 Sep;70(9):1064-76. doi: 10.1902/jop.1999.70.9.1064. PMID 10505810
- [Background] Huang LH, Neiva RE, Wang HL. Factors affecting the outcomes of coronally advanced flap root coverage procedure. J Periodontol. 2005 Oct;76(10):1729-34. doi: 10.1902/jop.2005.76.10.1729. PMID 16253095
- [Background] Cairo F, Rotundo R, Miller PD, Pini Prato GP. Root coverage esthetic score: a system to evaluate the esthetic outcome of the treatment of gingival recession through evaluation of clinical cases. J Periodontol. 2009 Apr;80(4):705-10. doi: 10.1902/jop.2009.080565. PMID 19335093